CLINICAL TRIAL: NCT02239029
Title: The Effect of Platelet Rich Plasma on Osteoarthritis of Knee
Brief Title: Platelet Rich Plasma on Osteoarthritis of Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yung-Tsan Wu (Other)
Responsible Party: Sponsor-Investigator, Yung-Tsan Wu, Attending Physician, Tri-Service General Hospital
Organization: Tri-Service General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSGHIRB-2-103-05-075; TSGHIRB-2-103-05-075, Taiwan (Other Grant/Funding Number: TSGHIRB-2-103-05-075, Taiwan)
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Knee Osteoarthritis
Keywords: Platelet rich plasma; Osteoarthritis of knee; Balance; Strength
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet rich plasma (Active Comparator): Platelet rich plasma (PRP) is a new and potential treatment for patients with kinds of musculoskeletal disorders.
  Patients with bilaetral knee osteoarthritis randomized receive on dose of PRP in one knee and placebo with normal saline in the other side.
  Interventions: Drug: platelet rich plasma
- normal saline (Placebo Comparator): Normal saline was injected into the other side of knee as the control group.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: platelet rich plasma — Platelet rich plasma (PRP) is a new and potential treatment for patients with kinds of musculoskeletal disorders.
  Arms: Platelet rich plasma
Drug: Normal saline — The normal salin as the placebo intervention was injection in the other side of knee.
  Arms: normal saline

SUMMARY:
Although few studies have showed beneficial effect of platelet rich plasma (PRP) for osteoarthritis of knee (OA knee), only one study applied randomized, control method and none of them has the objective measurements such as balance test or muscle strength which were reported as decrease in patients with OA knees. We assess the analgesic effect and the extent of improved muscle strength and balance after PRP in patients with OA knee.

DETAILED DESCRIPTION:
Patients with bilateral OA knee will be enrolled and randomized into intervention and control knee. One dose of PRP is applied in the intervention knee and normal saline in control side. Outcome measurements included visual analog scale (VAS)、Lequesne's severity index、Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)、balance test (Biodex) and isokinetic strengthening test at different follow-up frame (2nd week, 1st month, 3rd month and 6th month after treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 35 to 75 y/o.
2. Alert consciousness
3. Symptom of knee osteoarthritis persist at least 6 months and stage I or II scored by Ahlbäck grading system
4. The pain score measured by VAS at least 4 points

Exclusion Criteria:

1. Has received hyaluronic acid or steroid injection within 6 monts
2. Has received NSAIDs or steroid within one week
3. Tumor or metastasis surrounding the knee joint
4. Has received total knee replacement, major surgery in knee, rheumatoid arthritis
5. Patient who cant tolerance the balance or muscle strength test.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain on 2nd week, 1st month, 3rd month and 6th month after PRP. | Pre-treatment, 2nd week, 1st month, 3rd month and 6th month after PRP.
  Using the Visual analog scale (VAS) to measure the pain scale before treatment and multiple time frame after treatment.

SECONDARY OUTCOMES:
Change from baseline in severity of symptoms and functional status on 2nd week, 1st month, 3rd month and 6th month after treatment. | Pre-treatment, on 2nd week, 1st month, 3rd month and 6th month after treatment..
  Using the Lequesne's severity index to measure the symptoms and functional status before treatment and multiple time frame after treatment.
Change from baseline in severity of symptoms and functional status on 2nd week, 1st month, 3rd month and 6th month after treatment. | Pre-treatment and 2nd week, 1st month, 3rd month and 6th month after treatment.
  Using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) to measure the symptoms and functional status before treatment and multiple time frame after treatment.
Change from baseline in balance function on 2nd week, 1st month, 3rd month and 6th month after treatment. | Pre-treatment, 2nd week, 1st month, 3rd month and 6th month after treatment.
  Using the balance test (Biodex) to measure the balance function before treatment and multiple time frame after treatment.
Change from baseline in muscle strength of lower extremities on 2nd week, 1st month, 3rd month and 6th month after treatment. | Pre-treatment, 2nd week, 1st month, 3rd month and 6th month after treatment.
  Using the isokinetic strengthening test to measure the muscle strength of lower extremities before treatment and multiple time frame after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Cheng Chen, MD, MS, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, National Defense Medical Center
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center,, Taipei, Neihu District, Taiwan

REFERENCES:
- [Result] Matava MJ. Platelet-rich plasma: the next big thing?: commentary on an article by Ujash Sheth, BHSc, et al.: "Efficacy of autologous platelet-rich plasma use for orthopaedic indications: a meta-analysis". J Bone Joint Surg Am. 2012 Feb 15;94(4):e25. doi: 10.2106/JBJS.K.01423. No abstract available. PMID 22241605
- [Result] Patel S, Dhillon MS, Aggarwal S, Marwaha N, Jain A. Treatment with platelet-rich plasma is more effective than placebo for knee osteoarthritis: a prospective, double-blind, randomized trial. Am J Sports Med. 2013 Feb;41(2):356-64. doi: 10.1177/0363546512471299. Epub 2013 Jan 8. PMID 23299850
- [Result] Spakova T, Rosocha J, Lacko M, Harvanova D, Gharaibeh A. Treatment of knee joint osteoarthritis with autologous platelet-rich plasma in comparison with hyaluronic acid. Am J Phys Med Rehabil. 2012 May;91(5):411-7. doi: 10.1097/PHM.0b013e3182aab72. PMID 22513879
- [Result] Khalaj N, Abu Osman NA, Mokhtar AH, Mehdikhani M, Wan Abas WA. Balance and risk of fall in individuals with bilateral mild and moderate knee osteoarthritis. PLoS One. 2014 Mar 18;9(3):e92270. doi: 10.1371/journal.pone.0092270. eCollection 2014. PMID 24642715